CLINICAL TRIAL: NCT03347357
Title: Population Pharmacokinetics of Tacrolimus in Children With Nephrotic Syndrome
Brief Title: Pharmacokinetics of Tacrolimus in Children
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Wei Zhao, Head of department of clinical pharmacy and pharmacology, Shandong University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017TAC002
Record Dates: First submitted 2017-10-30; First posted 2017-11-20 (Actual); Last update posted 2017-11-20 (Actual); Status verified 2017-10

CONDITIONS: Nephrotic Syndrome
MeSH Terms: conditions — Nephrotic Syndrome | interventions — Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- tacrolimus (Experimental)
  Interventions: Drug: Tacrolimus

INTERVENTIONS:
Drug: Tacrolimus — Tacrolimus was administered orally at a dose of 0.05 mg/kg/dose twice daily (bid) for children with nephrotic syndrome.

SUMMARY:
the present study was conducted to assess the population pharmacokinetics of tacrolimus in children with nephrotic syndrome and to use these data to calculate an optimal dosing regimen of tacrolimus for use in these patients.

ELIGIBILITY:
Inclusion Criteria:

* patients have been diagnosed with nephrotic syndrome;
* age range: 1 month to 18 years old
* tacrolimus used as part of regular treatment

Exclusion Criteria:

* expected survival time less than the treatment cycle;
* patients with other factors that researcher considers unsuitable for inclusion.

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 28 (Actual)
Dates: Start 2012-01-01 (Actual); Primary Completion 2017-09-30 (Actual); Study Completion 2017-09-30 (Actual)

PRIMARY OUTCOMES:
change of plasma concentration of Tacrolimus | at 1,2,3,6,9,12 hours after oral administration
  To detect the plasma concentrations of Tacrolimus after oral administration

CONTACTS AND LOCATIONS:
Overall Officials: Wei Zhao, Ph.D, Principal Investigator — Shandong University